CLINICAL TRIAL: NCT00941564
Title: "Comparative Calcium Absorption and Gastrointestinal Tolerance in Healthy Term Infants Fed Milk-based Formulas With Different Fat Blends"
Brief Title: Comparative Ca Absorption and Tolerance in Healthy Term Infants Fed Milk-based Formulas With Different Fat Blends
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AK76
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Infant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Commercially available infant formula A (Experimental): Varying fat blend from comparator product
  Interventions: Other: Infant Formula milk based
- Commercially available infant formula B (Active Comparator)
  Interventions: Other: Infant formula milk based

INTERVENTIONS:
Other: Infant Formula milk based — Consume ad lib
  Arms: Commercially available infant formula A
Other: Infant formula milk based — consume ad lib
  Arms: Commercially available infant formula B

SUMMARY:
The objective is to assess the comparative calcium absorption and gastrointestinal (GI) tolerance in healthy normal term infants fed two commercially available powdered milk-based formulas which contain different fat blends.

ELIGIBILITY:
Inclusion Criteria:

* Infant in good health, full term, singleton birth and 84-156 days of age at enrollment. Male infants only to be enrolled for primary variable measures.
* Restrict use of certain medications or home remedies, herbal preparations, probiotics or rehydration/intravenous (IV) fluids.

Exclusion Criteria:

* Adverse maternal, fetal or infant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Infant has been treated with antibiotics 3 days prior to enrollment.
* Infant has received probiotics-containing products 3 days prior to enrollment.

Ages: 84 Days to 159 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Calcium absorption | 18 days

SECONDARY OUTCOMES:
Calcium retention, fat absorption, tolerance | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, PhD, Study Director — Abbott Nutrition
Locations (1):
- Department of Pediatrics, Federal University of Bahia, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Souza CO, Leite MEQ, Lasekan J, Baggs G, Pinho LS, Druzian JI, Ribeiro TCM, Mattos AP, Menezes-Filho JA, Costa-Ribeiro H. Milk protein-based formulas containing different oils affect fatty acids balance in term infants: A randomized blinded crossover clinical trial. Lipids Health Dis. 2017 Apr 14;16(1):78. doi: 10.1186/s12944-017-0457-y. PMID 28410612
- [Derived] Leite ME, Lasekan J, Baggs G, Ribeiro T, Menezes-Filho J, Pontes M, Druzian J, Barreto DL, de Souza CO, Mattos A, Costa-Ribeiro H Jr. Calcium and fat metabolic balance, and gastrointestinal tolerance in term infants fed milk-based formulas with and without palm olein and palm kernel oils: a randomized blinded crossover study. BMC Pediatr. 2013 Dec 24;13:215. doi: 10.1186/1471-2431-13-215. PMID 24367946